CLINICAL TRIAL: NCT02279160
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Phase 2 Trial of Ralinepag, an Oral IP Receptor Agonist, in Patients With Pulmonary Arterial Hypertension
Brief Title: Safety and Efficacy of APD811 in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APD811-003
Record Dates: First submitted 2014-10-25; First posted 2014-10-30 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ralinepag

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APD811 (Experimental): Multiple dose titration to maximum tolerated dose.
  Interventions: Drug: APD811
- Placebo (Placebo Comparator): Multiple dose titration to maximum tolerated dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD811
  Other Names: Ralinepag
  Arms: APD811
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study was conducted as a placebo-controlled, randomized, 22-week double-blind study which included a dose titration period. An additional transition period occurred for those patients who elected to enroll into the open-label extension study, APD811-007. A total of 61 patients with PAH were enrolled.

DETAILED DESCRIPTION:
Study APD811-003 was a 22-week, randomized, double-blind, parallel-group, placebo-controlled study in subjects with symptomatic WHO Group 1 PAH. The study consisted of a dose titration period of up to 9 weeks, a 13-week maintenance period, and a follow-up visit that was to occur approximately 3 weeks after the end of the maintenance period (Week 25). The transition period of 3 weeks (±1 week) was to occur for those subjects who elected to enroll into the open-label extension (OLE) Study APD811-007.

Approximately 60 subjects with PAH were planned to be enrolled (61 actual). After screening, eligible subjects were randomized 2:1 to ralinepag (APD811) or to placebo. Randomization was stratified by baseline WHO/NYHA functional class (II versus III or IV). Subjects randomized to active therapy were given ralinepag at a starting dose of 0.01 mg BID. Subjects randomized to the placebo arm received matching placebo capsules to preserve the blind. Subjects were instructed to take the study drug (ralinepag or placebo) with food. Dosage was then uptitrated, as tolerated, over the course of the 9-week dose-titration period to a maximum dose of 0.3 mg BID. Although doses could be reduced based on tolerability, the final dosage reached was required to be stable during the 13-week treatment period prior to evaluation at Week 22.

Subjects could receive concomitant oral disease-specific PAH therapy consisting of an ERA and/or an agent acting on the nitric oxide pathway, a PDE-5 inhibitor or a sGC stimulator, provided the dose had remained stable for at least 3 months prior to the start of screening. It was recommended that subjects continue the same dose and regimen of these medications for the duration of the study. With the exception of prostanoids, the use of other supporting therapies, which may affect PAH, was also permitted.

During the study, assessments of efficacy were performed including PVR and other hemodynamic parameters as determined by RHC, the 6MWT, assessment of clinical worsening, BNP and NT-proBNP levels, WHO/NYHA functional class assessment of PAH. Safety assessments included standard evaluations of AEs, clinical laboratory values, vital signs, and ECG measurements.

At the end of the maintenance period, subjects who did not choose to participate in the OLE study were to discontinue study drug (ralinepag or placebo). All subjects that chose to continue in the OLE study were to remain on study drug until the follow-up visit at Week 25. This visit served as the baseline visit for the OLE study if the subject was eligible and chose to participate.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-75 years, inclusive
* Symptomatic WHO Group 1 PAH classified by one of the following subgroups:

  * Idiopathic pulmonary arterial hypertension (IPAH);
  * Heritable pulmonary arterial hypertension (HPAH);
  * Drugs and toxins induced;
  * Associated pulmonary arterial hypertension (APAH); specifically connective tissue diseases, HIV infection and congenital heart disease.
* Has had the diagnosis of PAH confirmed by cardiac catheterization
* Has WHO/NYHA functional class II- IV symptomatology
* Previously diagnosed with PAH and on stable oral disease-specific PAH therapy with either an ERA and/or an agent acting on the nitric oxide pathway, i.e. a PDE5 inhibitor or a soluble guanylate cyclase stimulator. Stable is defined as no change in dose within 3 months of the start of Screening and for the duration of the study
* Has 6MWT distances of 100-500 m, and within 15% of each other on 2 consecutive tests done on different days at Screening
* Has pulmonary function tests (PFTs) within 6 months prior to the start of Screening with no evidence of significant parenchymal lung disease
* Has a ventilation-perfusion (V/Q) lung scan or pulmonary angiogram within 5 years prior to Screening and concomitant with or following diagnosis of PAH that shows no evidence of thromboembolic disease
* If on vasodilators (including calcium channel blockers), digoxin, spironolactone, or L-Arginine supplementation; the patient must be on a stable dose for at least 1 month prior to the start of Screening

Exclusion Criteria:

* Newly diagnosed with PAH and on no disease-specific PAH therapy
* Previous participation in any clinical study with an investigational drug, biologic, or device within 2 months prior to the Screening visit
* Acutely decompensated heart failure within 1 month prior to start of Screening
* Systolic blood pressure <90 mm Hg at Screening
* Evidence or history of left-sided heart disease and/or clinically significant cardiac disease
* Use or chronic administration (defined as >30 days) of a prostacyclin or prostacyclin analogue within 3 months of Screening
* Any previous use of a prostacyclin or prostacyclin analogue that was stopped for safety or tolerability issues associated with pharmacology/mechanism of action
* Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Solum, PhD, Study Director — United Therapeutics
Locations (35):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - UCLA Medical Center, Torrance, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - University of Texas, Houston Center for Clinical and Translational Sciences, Houston, Texas
- Australia (5):
  - The Prince Charles Hospital, Chermside
  - St Vincent's Hospital, Darlinghurst
  - St Vincent's Hospital, Fitzroy
  - Royal Hobart Hospital, Hobart
  - Fiona Stanley Hospital, Murdoch
- Bulgaria (2):
  - "Многопрофилната болница за активно лечение "Национална кардиологична болница "" ЕАД, Sofia
  - Многопрофилна болница за активно лечение "Света Анна" София АД, Клиника по кардиология, Sofia
- II. interní klinika - klinika kardiologie a angiologie, 1. lékařská fakulta, Univerzita Karlova v Praze a Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- Hungary (3):
  - Gottsegen György Országos Kardiologiai Intézet, Felnőtt Kardiológia, Budapest
  - Semmelweis Egyetem Pulmonológiai Klinika, Budapest
  - Pécsi Tudományegyetem Klinikai Központ, Szívgyógyászati Klinika, Pécs
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II w Krakowie, Krakow
  - Wojewódzki Szpital Specjalistyczny im. W. Biegańskiego w Łodzi, Lodz
- Romania (3):
  - Institutul de Urgență pentru Boli Cardiovasculare, Secția Clinică Cardiologie III, Bucharest
  - Institutul de Pneumoftiziologie "Marius Nasta", Secția Clinică Pneumoftiziologie IV, Bucharest
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie, Sectia Clinica Pneumologie II, Timișoara
- Serbia (3):
  - Klinički Centar Srbije (KCS), Klinika za kardiologiju, Belgrade
  - Kliničko-bolnički centar (KBC) Zemun,Klinika za internu medicinu,Sluzba kardiologije, Belgrade
  - Institut za plućne bolesti Vojvodine Sremska Kamenica (IPBVSK),, Kamenitz
- Spain (3):
  - Hospital Universitari General Vall d'Hebron, Servicio de Neumología, Barcelona
  - Hospital Clinic de Barcelona, Departamento de Pneumologia, Barcelona
  - Hospital 12 de Octubre, Departamento de Cardiologia, Madrid

REFERENCES:
- [Derived] Torres F, Farber H, Ristic A, McLaughlin V, Adams J, Zhang J, Klassen P, Shanahan W, Grundy J, Hoffmann I, Cabell C, Escribano Subias P, Sood N, Keogh A, D'Souza G, Rubin L. Efficacy and safety of ralinepag, a novel oral IP agonist, in PAH patients on mono or dual background therapy: results from a phase 2 randomised, parallel group, placebo-controlled trial. Eur Respir J. 2019 Oct 10;54(4):1901030. doi: 10.1183/13993003.01030-2019. Print 2019 Oct. PMID 31391223

RESULTS

PARTICIPANT FLOW:
Groups:
- APD811: Multiple dose titration to maximum tolerated dose.
  APD811
Period: Overall Study
Arm/Group | APD811 | Placebo
Started | 40 | 21
Completed | 34 | 19
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APD811 | Placebo | Total
Number analyzed (Participants) | 40 | 21 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 18 | 57
  >=65 years | 1 | 3 | 4
Age, Continuous [Median (Full Range); unit: years] | 46.5 [19 to 68] | 60 [29 to 73] | 51 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 38 | 19 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 38 | 19 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 4 | 10
  Bulgaria | 2 | 0 | 2
  Czechia | 3 | 1 | 4
  Hungary | 0 | 3 | 3
  Poland | 1 | 3 | 4
  Romania | 3 | 3 | 6
  Serbia | 8 | 3 | 11
  Spain | 7 | 2 | 9
  United States | 10 | 2 | 12
Weight [Median (Full Range); unit: kg] | 73.5 [43 to 122] | 68 [51 to 92] | 72.5 [43 to 122]
Height [Median (Full Range); unit: cm] | 160.5 [145 to 182] | 162 [145 to 170] | 161 [145 to 182]
BMI [Median (Full Range); unit: kg/m^2] | 27.18 [18.1 to 43.8] | 25.68 [19.4 to 38.3] | 27.13 [18.1 to 43.8]
Duration of PAH (Years) [Median (Full Range); unit: years] | 2.22 [0.3 to 27] | 1.76 [0.3 to 14] | 2 [0.3 to 27]
PAH Treatment [Count of Participants; unit: Participants]
  Monotherapy (ERA or PDE5-Inhibitor) | 14 | 11 | 25
  Combination Therapy (ERA + PDE5-Inhibitor/sGCS) | 26 | 10 | 36
PAH Classification [Count of Participants; unit: Participants]
  Idiopathic PAH | 21 | 11 | 32
  Heritable PAH | 4 | 1 | 5
  Drugs or Toxin Induced | 4 | 0 | 4
  Associated PAH | 11 | 9 | 20
Baseline WHO/NYHA Functional Class [Count of Participants; unit: Participants] — WHO FC I describes patients who do not experience symptoms with exercise or at rest. WHO FC II describes patients who experience symptoms with ordinary activities but not at rest. WHO FC III describes patients who are limited in normal activities but do not experience symptoms at rest. WHO FC IV describes patients who are symptomatic at rest and experience severe symptoms with any activity.
  Participants
    Class I | 0 | 0 | 0
    Class II | 22 | 12 | 34
    Class III | 17 | 9 | 26
    Class IV | 1 | 0 | 1
Baseline Pulmonary Vascular Resistance [Median (Full Range); unit: dyn*sec/cm^-5] | 704.6 [300 to 2119.4] | 479.7 [282.4 to 1600] | 575.7 [282.4 to 2119.4]
Baseline 6MWD [Median (Full Range); unit: meters] — The 6MWD is used to evaluate exercise capacity associated with carrying out activities of daily living. The 6-minute walk test (6MWT) should be administered by the same tester/on the same course at each site throughout the study. The area used for the 6MWT should be premeasured at approximately 30 m in length (but no shorter than 15 m [16 yards or 50 feet] in length at minimum) and at least 2 to 3 m in width. There should be no turns or curves. The length should be marked with gradations at least every 3 meters to ensure the accurate measurement of the distance walked.
  meters | 405 [105 to 686] | 367 [154 to 543] | 400 [105 to 686]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR)
Description: Measurements of PVR from right heart catheterization were obtained prior to Day 1 of the dose titration period and at the end of the maintenance period (Week 22), approximately 4 hours after the last dose of study drug.
Time Frame: Baseline and 22 Weeks
Population: Intent-to-Treat Population
Measure: Geometric Mean (Standard Deviation); unit: dyn*sec/cm^5
Arm/Group | APD811 | Placebo
Number analyzed (Participants) | 40 | 21
dyn*sec/cm^5 | 514.6 (1.85) | 512.0 (1.62)
Statistical Analysis 1: Comparison: APD811 vs Placebo; Test type: Superiority; p = 0.0220, ANCOVA; Multiple imputation = 0.742, 95% CI 2-sided [0.575 to 0.958]

2. Primary Outcome: Change From Baseline in 6-minute Walk Distance (6MWD) in Patients With PAH
Description: The 6MWT was conducted according to the modified guidelines issued by the American Thoracic Society prior to Day 1 of the dose titration period and at the end of the maintenance period (Week 22).
Time Frame: Baseline and 22 Weeks
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | APD811 | Placebo
Number analyzed (Participants) | 38 | 21
meters | 36.2 (11.79) | 29.4 (16.16)
Statistical Analysis 1: Comparison: APD811 vs Placebo; Test type: Superiority; p = 0.9002, Stratified Wilcoxon; Hodges-Lehmann estimate = 0.0, 95% CI 2-sided [-28.0 to 30.0]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time the subject provided informed consent through the duration of the study (up to 22 weeks).
Description: Adverse events were elicited at the time indicated in the schedule by asking the question: "Since you were last asked, have you felt unwell or different from usual in any way?" Any adverse or unexpected events, signs and symptoms were fully recorded on the Adverse Event form including details of intensity, onset, duration, outcome and relationship to the drug as determined by the PI.
Arm/Group | APD811 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 2/21
Serious Adverse Events (participants affected / at risk) | 4/40 | 6/21
Other Adverse Events (participants affected / at risk) | 40/40 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APD811 (N=40) | Placebo (N=21)
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APD811 (N=40) | Placebo (N=21)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Headache (Nervous system disorders) | 31 | 6
Nausea (Gastrointestinal disorders) | 20 | 5
Diarrhoea (Gastrointestinal disorders) | 19 | 3
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 14 | 3
Flushing (Vascular disorders) | 13 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 1
Vomiting (Gastrointestinal disorders) | 10 | 3
Abdominal Pain (Gastrointestinal disorders) | 7 | 0
Dizziness (Nervous system disorders) | 7 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Oedema peripheral (General disorders) | 6 | 1
Arthralgia (Metabolism and nutrition disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Urinary tract infection (Infections and infestations) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Influenza (Infections and infestations) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02279160/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02279160/SAP_001.pdf